CLINICAL TRIAL: NCT05899465
Title: Perioperative Treatment With Tranexamic Acid in Melanoma; Prognostic and Treatment-related Impact of the Plasminogen-plasmin Pathway
Brief Title: Perioperative Treatment With Tranexamic Acid in Melanoma
Acronym: PRIME
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRIME
Record Dates: First submitted 2023-04-04; First posted 2023-06-12 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Melanoma
Keywords: Melanoma; Tranexamic acid; Relapse; Cancer; Drug Repositioning; Surgery
MeSH Terms: conditions — Melanoma; Recurrence; Neoplasms | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel, two-arm, randomized, blinded Danish multi-center trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators/outcome assessors are all blinded to the intervention. Selected trained personnel who does not treat or assess the participants will be unblinded to prepare the intervention for administration and deliver the intervention to blinded personnel for administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid (Experimental): A single dose of TXA (15 mg/kg) administered intravenously 30 min (+/-15 min) before skin incision and subsequently, TXA (1000 mg) administered orally 4 and 8 hours post-surgery and TXA (1000 mg) 3 times daily through postoperative day 4.
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): A single dose of saline matching the volume of the experimental arm treatment regiment (Saline) administered intravenously 30 min (+/-15 min) before skin incision and subsequently, placebo tablets (2 tabs.) administered orally 4 and 8 hours post-surgery and (2 tabs) 3 times daily through postoperative day 4.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tranexamic acid — A single preoperative intravenous dose and per os treatment postoperatively day 1 through 4
  Arms: Tranexamic Acid
Drug: Saline — A single preoperative intravenous dose and per os treatment postoperatively day 1 through 4
  Arms: Placebo

SUMMARY:
Surgery is a key element in the treatment of melanoma, and naturally linked with an inflammatory response and recruitment of innate immune cells. Although surgery has a favorable intent, surgery-induced inflammation, neutrophils in particular, may accelerate growth of local and systemic micrometastases. Thus, improving cancer surgery and modulating the wound microenvironment in ways that benefit the patients is crucial.

Repurposing already approved drugs in a cancer setting has gained increasing interest in recent years. Interestingly, tranexamic acid was recently suggested as an anti-cancer drug, capable of reducing tumor growth in experimental animal models and reducing the viability of different melanoma cell lines.

As a novel approach, sponsor and investigators will conduct a Randomised Clinical Trial, using perioperative treatment with Tranexamic Acid, aiming to prevent the early relapses for patients with melanoma.

DETAILED DESCRIPTION:
The objective of the proposed clinical trial is to test if perioperative treatment with tranexamic acid (TXA) reduces the early relapses and postoperative complications for patients with melanoma and evaluate perioperative inflammation and the prognostic- and treatment-related impact of the plasminogen-plasmin pathway from human blood- and tissue samples.

Primary aim:

To test if perioperative treatment with TXA is superior to placebo and reduces the early relapse rates, from 37% to 26%, for patients diagnosed with melanoma undergoing sentinel lymph node biopsy surgery.

Secondary aims:

1. Evaluate safety and tolerability: defined as mild (abdominal pain, diarrhea, or nausea) or severe (thromboembolic events) adverse effects.
2. Evaluate postoperative complications: defined as bleeding, seroma formation, and infections within the first three postoperative months.
3. Estimate melanoma-specific survival probabilities and compare the two treatment groups.

Explorative:

From blood- and tissue samples, baseline and perioperative changes of factors associated with inflammation, fibrinolysis, metabolism, immune cell composition, and activation status will be monitored and factors will be associated with prognostic and treatment-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Diagnosed with invasive cutaneous melanoma (pathological stage/tumor grade ≥T2b), defined as either: Breslow thickness >1.0-2.0 mm with presence of ulceration or Breslow thickness >2.0 mm regardless of ulceration status.
* Eligible for surgery (wide local excision and sentinel lymph node biopsy).
* >/=18 years of age and </=80 years of age
* Signed Informed Consent Form

Exclusion Criteria:

Patients

* With a prior history of invasive melanoma
* Thromboembolic events within the last 3 months
* Pregnancy
* Active breastfeeding
* Known allergy or hypersensitivity to TXA
* Known and treated epilepsia or previous seizures
* eGFR 0-50
* Current use of tranexamic acid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1204 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in rate of relapse within two years when comparing treatment arms | 2 year follow-up
  Histopathological confirmed relapse, defined as either local, regional (in transit or lymph node) or systemic relapses. Systemic metastases suspected on PET / CT/ MR will be used if a biopsy is not possible. Based on the primary endpoint, we will calculate the relapse risk proportions for each treatment arm as a binary outcome.
  The date of relapse or completed follow-up is noted and the relapse-free period is defined as the date of wide local excision and sentinel lymph node biopsy until the date of either the first confirmed relapse or the date of completed two-year follow-up without relapse.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events | 6 months follow-up
  Adverse events summarised according to grade:
  Mild: defined as the patient's report of abdominal pain, diarrhea, or nausea. Severe: thromboembolic events, verified radiologically.
Assessment of incidens of postoperative complications | 3 months follow-up
  Postoperative complications, summarised according to the type and postoperative timepoint, is defined as binary outcomes:
  Bleeding: defined as a drained or surgically removed hematoma or suggillation of blood to the skin around the operated area, occurring within the first 10 days post-surgery.
  Seroma: drained seroma, during the period from end of surgery through 3 months post-surgery.
  Infection: local wound infection, treated with antibiotics or surgical intervention, during the period from end of surgery through 3 months post-surgery.
Melanoma-specific survival | 2 year follow-up
  Time to event estimates:
  Defined as the period from the date of surgery (wide local excision and sentinel lymph node biopsy) to the date of death from suspected systemic melanoma (histopathologically confirmed relapse or systemic metastases suspected on PET / CT / MR) or the date of completed 2 years follow-up.
Overall survival | 2 year follow-up
  Time to event estimates:
  Defined as the period from the date of surgery (re-excision and sentinel node) to the date of death from all causes or the date of finalised 2 years follow-up.
Relapse free survival | 2 year follow-up
  Time to event estimates:
  Defined as the period from the date of surgery (re-excision and sentinel node) to the date of histopathologically confirmed relapse (local, regional or systemic), death from all causes or the data or completed 2 years follow-up.

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Aarhus University Hospital. Dept. of Plastic- and Breast Surgery, Aarhus, Central Jutland
  - Aalborg University Hospital. Dept. of Plastic- and Breast Surgery., Aalborg, North Denmark
  - Copgenhagen University Hospital, Rigshospitalet. Dept. of Plastic Surgery and Burns Treatment, Copenhagen
  - Copenhagen University Hospital, Herlev. Dept. of Plastic Surgery, Herlev
  - Sygehus Lillebælt, Vejle Hospital. Dept. of Plastic Surgery, Vejle

IPD SHARING:
Plan to Share IPD: Yes
Entirely anonymized data will be shared only upon reasonable request made to the sponsor and evaluated by the steering committee. Researchers requesting access are required to sign a data access agreement assuring that data will only be utilized for a predetermined and accepted purpose.
Supporting Information: Study Protocol, SAP, ICF
URL: https://www.ema.europa.eu/en

REFERENCES:
- [Derived] Kristjansen KA, Engel Krag A, Schmidt H, Holmich LR, Bonnelykke-Behrndtz ML. Perioperative treatment with tranexamic acid in melanoma (PRIME): protocol for a Danish multicentre randomised controlled trial investigating the prognostic and treatment-related impact of the plasminogen-plasmin pathway. BMJ Open. 2024 Feb 2;14(2):e077012. doi: 10.1136/bmjopen-2023-077012. PMID 38309757